CLINICAL TRIAL: NCT06005545
Title: A Comparative Evaluation of Effectiveness in Root Canal Debridement Using Inertial Cavitation Device vs Passive Ultrasonic Irrigation and Conventional Preparation: A Randomized Controlled Clinical Trial
Brief Title: A Study to Compare Various Root Canal Cleaning Devices Based on Cavitation,Ultrasonic and Conventional Methods.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lumendo AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC_5301_V1.0_CIP
Record Dates: First submitted 2023-08-08; First posted 2023-08-22 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Apical Periodontitis
Keywords: Root Canal Treatment; Endodontic Treatment; Root Canal Debridement
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: This is a prospective, 3- arm randomized, non-blinded, single center pivotal clinical investigation, performed to evaluate the effectiveness and safety of the Endoclean device with 2 comparator arms.
  Arm 1: Passive ultrasonic irrigation group (PUI); shaping up to WL with 25.06, Arm 2: Endoclean (EC) group; shaping up to WL with 20.06; EC application tip kept 3mm short of WL, irrigation protocol with NaOCl (sodium hypochlorite) Arm 3: Conventional group; shaping up to WL of 25.06, irrigation protocol with NaOCl (sodium hypochlorite)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Passive Ultrasonic Irrigation group (PUI) (Active Comparator): Arm 1: Passive ultrasonic irrigation group (PUI); shaping up to WL with 25.06,
  Interventions: Device: Passive Ultrasonic Irrigation (PUI) group
- Endoclean group (EC) (Experimental): Arm 2: Endoclean (EC) group; shaping up to WL with 20.06; EC application tip kept 3mm short of WL, irrigation protocol with NaOCl (sodium hypochlorite)
  Interventions: Device: Endoclean (EC) group
- Conventional Group (Active Comparator): Arm 3: Conventional group; shaping up to WL of 25.06, irrigation protocol with NaOCl (sodium hypochlorite)
  Interventions: Device: Conventional group

INTERVENTIONS:
Device: Passive Ultrasonic Irrigation (PUI) group — Passive ultrasonic irrigation is the current golden standard in root canal cleaning and irrigation devices. It is used after root canal shaping using manual or rotary instruments. It uses sodium hypochlorite which is mobilized in the canal using ultrasonic non-cutting tips to clean, debride, disinfect, and prepare the root canal for obturation.
  Other Names: Ultrasonic group
  Arms: Passive Ultrasonic Irrigation group (PUI)
Device: Endoclean (EC) group — Endoclean is a novel device that uses hydraulic inertial cavitation with the help of pressure and saline solution to debride the root canal after minimal shaping using manual or rotary shaping instruments. It is used to effectively clean, debride and prepare the root canal before obturation in the root canal treatment procedure.
  Other Names: Cavitation group
  Arms: Endoclean group (EC)
Device: Conventional group — Conventional root canal preparation uses manual or rotary files along with manual irrigation using syringes and irrigant solutions like sodium hypochlorite or EDTA to clean, debride and prepare the root canal for obturation.
  Arms: Conventional Group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of various root canal cleaning devices based on the principle of cavitation, ultrasonics, and conventional methods in a normal healthy adult population aged between 18 to 75 years requiring root canal treatment.

The main question[s] it aims to answer are:

* Effectiveness of the cleaning mechanism
* Evaluate the safety of use of the device. Participants will be provided root canal treatment. Participants will be asked to record their post-operative pain levels in a Patient Pain diary. The healing rate of the lesion will be examined at follow-up visits using intraoral X-rays. At the end of the study, a statistical analysis of the clinical outcomes of the root canal treatment will be examined and evaluated in every group.

DETAILED DESCRIPTION:
Study title: "A Comparative Evaluation of Effectiveness in Root Canal Debridement using Inertial Cavitation Device vs Passive Ultrasonic Irrigation and Conventional Preparation: A Randomized Controlled Clinical Trial".

Study Design: This is a prospective, 3-arm randomized, non-blinded, single-center pivotal clinical investigation, performed to evaluate the effectiveness and safety of the Endoclean device with 2 comparator arms.

Primary objective: To test the effectiveness of the Endoclean device for root canal debridement up to 12-month follow-up.

Secondary objective: To test the extended effectiveness and safety of the Endoclean device up to a 24-month follow-up.

Inclusion/Exclusion Criteria:

1. Inclusion Criteria

   •Patients aged between 18-75 years with ASA (American Society of Anesthesiologists) classification 1 and 2.

   ASA 1: A normal healthy patient. Example: Fit, non-obese BMI (Body mass index) under 30, a non-smoking patient with good exercise tolerance.

   ASA 2: A patient with mild systemic disease. Example: Patient with no functional limitations and a well-controlled disease (e.g., treated hypertension, obesity with BMI under 35, frequent social drinker, or cigarette smoker).
   * Patients who agreed to participate and who have signed the informed consent.
   * Patients presenting with symptomatic and/or asymptomatic apical periodontitis and radiographic evidence of apical periodontitis in anterior or posterior teeth larger than 1.5 mm in diameter.
   * Mature tooth with closed apices
   * Tooth that has never been treated with root canal therapy.
2. Exclusion Criteria:

   * Patients, who have pre-existing health or oral conditions that placed them at risk during the trial.
   * Patients with generalized untreated periodontal disease.
   * Patients with a history of analgesic intake within the past 3 days or antibiotics in the last 1 month.
   * Uncooperative patients
   * Teeth with immature apices, root resorption, or requiring extensive prosthetic rehabilitation.
   * Teeth that cannot be made functional nor restored or difficult to access teeth with no importance (wisdom teeth)
   * Teeth with insufficient periodontal support
   * Teeth with poor prognosis, for example due to deep root caries, large root resorption or open apex cases
   * Fractured teeth
   * Local anatomical factors such as an inaccessible root end
   * Presence of fractured instrument in the root canal
   * Pregnant women
   * Patients unable to understand the study procedure.

Number of Participants:

Total number of participants = 109 subjects Arm 1: 40 subjects Arm 2: 40 subjects Arm 3: 29 subjects Test device: Endoclean (Lumendo AG): hydraulic cavitation cleaning device Control device 1: Passive ultrasonic irrigation (PUI) Control device 2: Rotary files with standard NaOCl irrigation Study duration: 2-3 years The results of the Endoclean group shall be compared to data gathered from the comparator device groups and results shall be presented in the clinical investigation report.

ELIGIBILITY:
Inclusion Criteria:

•Patients aged between 18-75 years with ASA (American Society of Anesthesiologists) classification 1 and 2.

ASA 1: A normal healthy patient. Example: Fit, non-obese BMI (Body mass index) under 30, a non-smoking patient with good exercise tolerance.

ASA 2: A patient with mild systemic disease. Example: Patient with no functional limitations and a well-controlled disease (e.g., treated hypertension, obesity with BMI under 35, frequent social drinker, or cigarette smoker).

* Patients who agreed to participate and who have signed the informed consent.
* Patients presenting with symptomatic and/or asymptomatic apical periodontitis and radiographic evidence of apical periodontitis in anterior or posterior teeth larger than 1.5 mm in diameter.
* Mature tooth with closed apices
* Tooth that has never been treated with root canal therapy.

Exclusion Criteria:

* Patients, who have pre-existing health or oral conditions that placed them at risk during the trial.
* Patients with generalized untreated periodontal disease.
* Patients with a history of analgesic intake within the past 3 days or antibiotics in the last 1 month.
* Uncooperative patients
* Teeth with immature apices, root resorption, or requiring extensive prosthetic rehabilitation.
* Teeth that cannot be made functional nor restored or difficult to access teeth with no importance (wisdom teeth)
* Teeth with insufficient periodontal support
* Teeth with poor prognosis, for example due to deep root caries, large root resorption or open apex cases
* Fractured teeth
* Local anatomical factors such as an inaccessible root end.
* Presence of fractured instrument in the root canal
* Pregnant women
* Patients unable to understand the study procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness endpoint | 12 months
  Successful healing of periapical lesion up to 12 months post-procedure where success is defined as completely healed or healing lesion with absence of clinical symptoms.
  Healing is assessed by measuring the reduction in periapical lesion radiolucency, up to 12 months post-procedure, using the PAI (periapical index score).
  The absence of clinical symptoms is defined as:
  1. The patient had no discomfort in treated tooth
  2. The patient had no percussive pain during the examination in treated tooth

SECONDARY OUTCOMES:
Safety endpoint | 1 month
  Freedom from postoperative pain up to 7 days of follow-up period (24 hours, 48 hours, 72 hours, 7 days and 1 month). Pain is measured by Visual Analogue Scale (VAS) assessment.The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. It consists of a line, approximately 10-15 cm in length, with the left side signifying no pain with a smiling face image and the right side signifying the worst pain ever with a frowning face image. The VAS is used to assist individuals to determine pain levels, who may not be accustomed to rating their pain on other types of scales, such as a numeric rating scale.
Secondary effectiveness endpoints | 24 months
  Successful healing of periapical lesion up to 24 months post-procedure. Long-term effectiveness success shall be defined as a continued reduction or complete absence of periapical lesion radiolucency at 24m FU since the procedure with no clinical symptoms (i.e no discomfort in treated tooth and no percussive pain during examination)

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medipol Universitesi, Faculty of Dentistry, Department of Endodontics, Istanbul, Unkapanı, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No